CLINICAL TRIAL: NCT02787382
Title: Myocardial Screening in Fetuses With Congenital Cytomegalovirus (CMV) Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0804-15-TLV
Record Dates: First submitted 2016-02-18; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Disorder of Cardiac Function
Keywords: cytomegalovirus; TORCH; prenatal diagnosis; congenital infections; fetal abnormalities; echocardiography; myocardial deformation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnant women with CMV infection (Experimental): An attempt to record the fetal myocardium will be done at the initial examination and at all the follow up examinations performed during pregnancy (every 3-4 weeks according to the clinical protocol currently in use at the OB-GYN US Unit).
  The participants will undergo a detailed fetal echocardiography according to standard guidelines (see below, section echocardiography).
  Interventions: Device: echocardiographic examination
- Pregnant women with suspected CMV infection (Experimental): The healthy women from the group will serve as controls. An attempt to record the fetal myocardium will be done at the initial examination and at all the follow up examinations performed during pregnancy (every 3-4 weeks according to the clinical protocol currently in use at the OB-GYN US Unit).
  The participants will undergo a detailed fetal echocardiography according to standard guidelines (see below, section echocardiography). As the control group-Newborns found to be negative for CMV will serve as control group.
  Interventions: Device: echocardiographic examination

INTERVENTIONS:
Device: echocardiographic examination — Patients will undergo echocardiography (us) starting at the time of the first referral and every 3-4 weeks until delivery and at the 2-7th day birth. Cardiac scans of fifty pregnant women the healthy women from the group will serve as controls at the 2-7th day birth. Cardiac scans of fifty pregnant women and the healthy women from the group will serve as controls
  EXPECTED RESULTS Subtle myocardial deformation abnormalities are expected to be commonly found in fetuses and infants with CMV infection.

SUMMARY:
BACKGROUND

Myocarditis and pericarditis are inflammatory conditions of the heart commonly due to viral or autoimmune etiologies. Human CMV represents one of the leading causes of congenital infections worldwide. There is limited data regarding the cardiac function of fetuses and infants with CMV.

OBJECTIVE

To provide insight regarding the presence of myocardial involvement in fetuses and infants with CMV infection.

PATIENTS & METHODS

Up to 100 fetuses with suspected CMV infection will be enrolled during a 3 years period. Patients will undergo detailed US examinations including dedicated neurosonography and echocardiography starting at the time of the first referral and every 3-4 weeks until delivery and at the 2-7th day birth. Cardiac scans of fifty pregnant women and the healthy women from the group will serve as controls

DETAILED DESCRIPTION:
BACKGROUND

Myocarditis and pericarditis are inflammatory conditions of the heart commonly due to viral or autoimmune etiologies. Human CMV represents one of the leading causes of congenital infections worldwide. There is limited data regarding the cardiac function of fetuses and infants with CMV.

OBJECTIVE

To provide insight regarding the presence of myocardial involvement in fetuses and infants with CMV infection.

PATIENTS & METHODS

Up to 100 fetuses with suspected CMV infection will be enrolled during a 3 years period. Patients will undergo detailed US examinations including dedicated neurosonography and echocardiography starting at the time of the first referral and every 3-4 weeks until delivery and at the 2-7th day birth. Cardiac scans of fifty pregnant women and the healthy women from the group will serve as controls

EXPECTED RESULTS

Subtle myocardial deformation abnormalities are expected to be commonly found in fetuses and infants with CMV infection.

CONCLUSIONS

The findings of this present study will underscore the need for cardiac screening of fetuses and infants with congenital CMV infection, with long-term follow-up to document the natural history and disease burden of CMV in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred because of suspected CMV IUI as demonstrated by seroconversion during pregnancy or during the 3 months that precede LMP or
2. Patients referred because of suspected CMV IUI based on the presence borderline CMV serology
3. US signs indicative of intrauterine CMV infection (CNS and non CNS involvement).

Exclusion Criteria:

1. Multifetal pregnancy.
2. Pregnant women planning to deliver elsewhere who are offered yet refuse to participate in the postnatal investigation following discharge from the hospital.
3. Patients will be excluded if they had clinical heart failure, as defined by the New York Heart Association classification (NYHA, class II-IV) (Criteria committee of NYHA 1994), a history of cardiovascular disease or chronic renal insufficiency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
diastolic strain RATE | 5 month
  US test will measure diastolic strain RATE (will be measured by %)
systolic strain RATE | 5 month
  US test will measure systolic strain RATE (will be measured by %)

CONTACTS AND LOCATIONS:
Overall Officials: Livia kapusta, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No